CLINICAL TRIAL: NCT00454155
Title: A Phase I/II Study of the Safety and Pharmacokinetics of Opebacan (rBPI21) in Patients Undergoing Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Study of Opebacan in Patients Undergoing Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Acronym: HSCT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BPSC030
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2011-05

CONDITIONS: Graft Versus Host Disease
Keywords: HSCT; AGVHD; Myeloablative; Allogeneic; Hematopoietic; Stem; Cell; Transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Opebacan (Experimental)
  Interventions: Drug: Opebacan

INTERVENTIONS:
Drug: Opebacan — 4 mg/kg continuous IV infusion for 30 minutes followed immediately by 6 mg/kg/day continuous IV infusion for 3 days

SUMMARY:
The objectives of this study are as follows:

To demonstrate the safety of escalating doses of opebacan in subjects undergoing myeloablative allogeneic Hematopoietic Stem Cell Transplantation

To determine the pharmacokinetics of opebacan in subjects undergoing myeloablative allogeneic Hematopoietic Stem Cell Transplantation

To determine if IV administration of opebacan is associated with changes in biological markers for inflammation

To develop preliminary descriptive data on the occurrence and severity of Hematopoietic Stem Cell Transplantation related complications, including aGvHD

DETAILED DESCRIPTION:
IV infusion of opebacan to replace endogenous BPI during the peritransplant period will result in the reduction of LPS-induced inflammatory sequelae, in particular aGvHD, in patients undergoing allogeneic HSCT.

The rationale for using opebacan in patients undergoing myeloablative regimens and HSCT is based on the following:

Endotoxemia has been demonstrated to play a central pathophysiologic role as a trigger of aGvHD in animal models.

Endotoxemia following HSCT is associated with inflammatory conditions (such as inflammatory cytokine release) that have been demonstrated in humans to be associated with organ damage and increased morbidity and mortality.

Endotoxemia and LBP elevation have been demonstrated in humans undergoing ablative HSCT.

Chemotherapy-induced neutropenia results in a deficiency of endogenous BPI levels.

The timing of the endotoxemic insult is predictable (i.e., subsequent to myeloablative chemotherapy and radiotherapy).

The return to normal neutrophil levels is not immediate and takes one week to several weeks.

Well established laboratory techniques for surrogate markers related to LPS presence and its activities can facilitate the evaluation of molecules designed to inhibit or antagonize LPS and its effects.

The objectives of this study are as follows:

To demonstrate the safety of escalating doses of opebacan in subjects undergoing myeloablative allogeneic Hematopoietic Stem Cell Transplantation

To determine the pharmacokinetics of opebacan in subjects undergoing myeloablative allogeneic Hematopoietic Stem Cell Transplantation

To determine if IV administration of opebacan is associated with changes in biological markers for inflammation

To develop preliminary descriptive data on the occurrence and severity of Hematopoietic Stem Cell Transplantation related complications, including aGvHD

ELIGIBILITY:
Inclusion Criteria:

* Age <= 60 and undergoing allogeneic HSCT
* Life expectancy > 8 weeks
* Scheduled for treatment with a conditioning regimen intended to be myeloablative
* Female subjects of child-bearing age must have a negative urine pregnancy test. Sexually active male and female subjects of reproductive age must be using a form of contraception considered effective and medically acceptable by the Investigator.

Exclusion Criteria:

* Cumulative lifetime exposure of > 300 mg/M2 of anthracycline (expressed as doxorubicin equivalent dose) or receipt of anthracycline within 180 days prior to initiating conditioning for HSCT
* Active infection
* Prophylactic antibacterial antibiotics.
* Positive for HIV, HTLV-I, or HTLV-II
* Any prior stem cell transplant
* Prior history of CHF
* Cord blood is the source of a subject's transplanted cells.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Time to engraftment | 100 days
Inflammatory markers | 100 days
Inflammatory states | 100 days
Transplant-related complications | 100 days
The pharmacokinetics of opebacan | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Guinan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Boston, Massachusetts, United States